CLINICAL TRIAL: NCT07036991
Title: A Randomized Clinical TRial on Inhibitor of PCSK9 and Statin Treatment for Carotid Artery Stenosis (TRIP-CAS)
Brief Title: Clinical Trial of PCSK9 Inhibitor and Statin Treatment for Carotid Artery Stenosis
Acronym: TRIP-CAS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRIP-CAS
Record Dates: First submitted 2025-05-29; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Carotid Artery Stenosis
Keywords: CAS; Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — evolocumab; Rosuvastatin Calcium; liptruzet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCSK9 Inhibitor + Statin ± Ezetimibe Group (Experimental): PCSK9 inhibitor (biweekly injections) + rosuvastatin/atorvastatin ± ezetimibe, initiated on randomization day
  Interventions: Drug: Evolocumab (biweekly injections) + Rosuvastatin/Atorvastatin ± Ezetimibe
- Statin ± Ezetimibe Group (Active Comparator): Rosuvastatin/atorvastatin ± ezetimibe, continued or initiated on randomization day
  Interventions: Drug: Rosuvastatin/Atorvastatin ± Ezetimibe

INTERVENTIONS:
Drug: Evolocumab (biweekly injections) + Rosuvastatin/Atorvastatin ± Ezetimibe — PCSK9 inhibitor (biweekly injections) + rosuvastatin/atorvastatin ± ezetimibe
  Arms: PCSK9 Inhibitor + Statin ± Ezetimibe Group
Drug: Rosuvastatin/Atorvastatin ± Ezetimibe — Rosuvastatin/atorvastatin ± ezetimibe
  Arms: Statin ± Ezetimibe Group

SUMMARY:
A prospective, multicenter, randomized controlled, open-label, blinded outcome evaluation (PROBE) trial.

DETAILED DESCRIPTION:
The trial is to evaluate the effect of ultra-intensive lipid-lowering therapy (PCSK9 inhibitor + rosuvastatin or atorvastatin, with/without ezetimibe) versus conventional lipid-lowering therapy (rosuvastatin or atorvastatin, with/without ezetimibe) on changes in atherosclerotic burden in patients with carotid artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria:

1. Age ≥ 18 years.
2. Asymptomatic mild-to-moderate carotid artery stenosis confirmed by CTA, MRA, ultrasound, or DSA, with no anticipated need for surgical intervention.
3. Modified Rankin Scale (mRS) score ≤ 2
4. Signed informed consent form obtained from the subject

Ultrasound Inclusion Criteria:

Carotid ultrasound showing a plaque burden rate ≥30% at the most stenotic cross-sectional site of the carotid artery (common carotid artery or proximal C1 segment of the internal carotid artery).

Exclusion Criteria:

1. Non-atherosclerotic carotid stenosis, including arterial dissection, Takayasu arteritis, radiation-induced vasculopathy, fibromuscular dysplasia, neurofibromatosis, suspected vasospasm, or recanalized vascular embolism.
2. Known cardioembolic sources: mitral stenosis, mechanical heart valve, infective endocarditis, intracardiac thrombus/vegetation, myocardial infarction within 3 months, dilated cardiomyopathy, chronic/paroxysmal atrial fibrillation. (Confound ASCVD outcome assessment.)
3. History of cerebrovascular, coronary, or peripheral arterial endovascular intervention within 30 days before enrollment or anticipated surgery within the next 6 months.
4. History of ischemic stroke, transient ischemic attack (TIA), or intracranial hemorrhage (parenchymal, subarachnoid, subdural, or epidural) before enrollment.
5. Pre-existing intracranial tumor, cerebral aneurysm, or arteriovenous malformation.
6. History of thromboembolic diseases (pulmonary embolism, mesenteric embolism, lower limb arterial embolism) or coronary atherosclerotic heart disease.
7. Severe neurological deficits impairing independent living; diagnosed dementia/psychiatric disorders interfering with follow-up; or life expectancy <3 years due to other conditions.
8. Severe/unstable comorbidities: Severe heart failure (NYHA Class III/IV or LVEF <30%), Renal failure (serum creatinine >264 μmol/L or creatinine clearance <0.6 mL/s), Severe hepatic dysfunction (ALT/AST >3× upper limit of normal), CK >5× upper limit of normal, Active malignancy.
9. Use of PCSK9 inhibitors or CETP inhibitors within 24 weeks before enrollment.
10. The subjects have taken strong inhibitor drugs of cytochrome P-450 3A4 (including: adagrasib, atazanavir, ceritinib, clarithromycin, darunavir, idelalisib, indinavir, itraconazole, ketoconazole, levonorgestrel, lonafarnib, lopinavir, mifepristone, nefazodone, nelfinavir, nirmatrelvir/ritonavir, Viekira Pak (ombitasvir, paritaprevir, and ritonavir tablets), mbitasvir/paritaprevir/ritonavir and dasabuvir, posaconazole, co-formulations containing ritonavir and ritonavir itself, saquinavir, erythromycin, tucatinib, voriconazole) within one month before randomization, or may require such drugs during the study period.
11. Pregnancy or lactation.
12. Concurrent participation in another trial that may affect outcome assessment.
13. Other situations that the investigator believes may cause significant harm to the subjects if they participate in this trial.
14. Situations where the investigator believes there are other vascular lesions that may lead to short - term ischemic events and surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in plaque burden rate at the most stenotic carotid site at 180±7 days | 180±7 days

SECONDARY OUTCOMES:
Lipid profile (TG/TC/LDL-C/HDL-C), liver function (ALT, AST), CK, CRP at 30±3 days | 30±3 days
Lipid profile (TG/TC/LDL-C/HDL-C/Lp(a)/ApoA1/ApoB), liver function (ALT, AST), CK, CRP at 90±3 days | 90±3 days
Carotid plaque burden rate at 90±3 days | 90±3 days
Carotid plaque diameter stenosis at 90±3 days | 90±3 days
Carotid plaque dimensions (length × thickness) at 90±3 days | 90±3 days
Plaque stability (hypoechoic regions, fibrous cap integrity, ulceration, plaque score) at 90±3 days | 90±3 days
Lipid profile: TG/TC/LDL-C/HDL-C/Lp-a/ApoA1, ApoB; liver function: ALT, AST, CK, CRP at 180±7 days | 180±7 days
Plaque burden rate at the most stenotic cross-sectional site of the carotid artery at 180±7 days | 180±7 days
Plaque diameter stenosis at 180±7 days | 180±7 days
Plaque dimensions (length × thickness) at 180±7 days | 180±7 days
Plaque stability (hypoechoic regions, fibrous cap integrity, ulceration, plaque score) at 180±7 days | 180±7 days
mRS score at 180±7 days | 180±7 days
Time to first major vascular event within 180±7 days (stroke/TIA, angina, myocardial infarction, symptomatic peripheral vascular disease) | within 180±7 days
mRS score at 365±30 days | 365±30 days
Time to first major vascular event within 365±30 days (stroke/TIA, angina, myocardial infarction, symptomatic peripheral vascular disease) | within 365±30 days

OTHER OUTCOMES:
Deaths within 180±7 days after enrolment | within 180±7 days after enrolment
SAEs within 180±7 days after enrolment | within 180±7 days after enrolment
ALT/AST >2× upper limit, CK >3× upper limit within 180±7 days after enrolment | within 180±7 days after enrolment
Deaths within 365±30 days after enrolment | within 365±30 days after enrolment
SAEs within 365±30 days after enrolment | within 365±30 days after enrolment
ALT/AST >2× upper limit, CK >3× upper limit within 365±30 days after enrolment | within 365±30 days after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital; Pinjing Hui, MD, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: Yes
Researchers need to submit a formal data sharing application to the TRIP-CAS Steering Committee and obtain the approval of the Steering Committee.
Supporting Information: Study Protocol, SAP
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research. 4.Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5.The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses.
URL: https://www.ocin.org.cn/